CLINICAL TRIAL: NCT00550225
Title: A Randomised, Double-blind, Dose Escalating Study in Healthy Volunteers to Assess the Safety, Tolerability, Extra Pulmonary Pharmacodynamics and Pharmacokinetics of Single Doses of GSK961081 (Succinate Salt)
Brief Title: Succinate Salt Version of GSK961081 for Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: MAB108115
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: succinate; anti-muscarinic; b-agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sequence 1 (Experimental): In session 1, subjects will receive 300 microgram GSK961081 succinate followed by placebo in session 2. The subjects will receive 1500 micrograms of GSK961081 succinate in session 3 and 1500 micrograms of GSK961081 edisylate in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 2 (Experimental): In session 1, subjects will receive 300 microgram GSK961081 succinate followed by 1500 micrograms of GSK961081 edisylate in session 2. The subjects will receive 1500 micrograms of GSK961081 succinate in session 3 and placebo in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 3 (Experimental): In session 1, subjects will receive 300 microgram GSK961081 succinate followed by placebo in session 2. The subjects will receive 1500 micrograms of GSK961081edisylate in session 3 and an additional dose of GSK961081 succinate in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 4 (Experimental): In session 1, subjects will receive 300 microgram GSK961081 succinate followed by 1500 micrograms of GSK961081 edisylate in session 2. The subjects will receive placebo in session 3 and an additional dose of GSK961081 succinate in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 5 (Experimental): In session 1, subjects will receive 1500 micrograms of GSK961081 edisylate followed by 900 microgram GSK961081 succinate in session 2. The subjects will receive 1500 micrograms of GSK961081 succinate in session 3 and placebo in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 6 (Experimental): In session 1, subjects will receive placebo followed by 900 micrograms of GSK961081 succinate in session 2. The subjects will receive 1500 micrograms of GSK961081 succinate in session 3 and 1500 micrograms of GSK961081 edisylate in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 7 (Experimental): In session 1, subjects will receive 1500 micrograms of GSK961081 edisylate followed by 900 microgram GSK961081 succinate in session 2. The subjects will receive placebo in session 3 and an additional dose of GSK961081 succinate in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo
- Sequence 8 (Experimental): In session 1, subjects will receive placebo followed by 900 microgram GSK961081 succinate in session 2. The subjects will receive 1500 micrograms of GSK961081 edisylate in session 3 and an additional dose of GSK961081 succinate in session 4.
  Interventions: Drug: GSK961081; Drug: GSK961081 matching placebo

INTERVENTIONS:
Drug: GSK961081 — GSK961081 edisylate and succinate will be administered as capsules via DISKUS inhaler formulated with lactose as a vehicle to make 12.5 milligrams. GSK961081 succinate will be given in a dose-ascending manner with a starting dose of 300 micrograms. The dose of GSK961081 edisylate is 1500 micrograms.
Drug: GSK961081 matching placebo — GSK961081 matching placebo formulated with lactose only as a vehicle to 12.5 milligrams will be administered via the DISKUS inhaler.

SUMMARY:
Salt Bridging study for GSK961081

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or female aged between 18 and 50 years.
* Body mass index within the range 19-29.9 kilograms/metre2
* Forced Expiratory Volume in 1 second (FEV1) >80% predicted and a FEV1/ Forced Vital Capacity (FVC) ratio > 0.7
* Subjects are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of < 10 pack years.

Exclusion criteria:

* Who have a past or present disease, which as judged by the Investigator and medical monitor may affect the outcome of the study or the safety of the subject
* History of respiratory disease
* Significant abnormal 12 lead ECG, QTc(B) and QTc(F) value at screening >450msec on an individual ECG or a PR interval outside the range 120-210 msec
* Supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* Subject has donated a unit of blood within the 56 days or intends to donate within 56 days after completing the study
* Subject is currently taking regular (or course of) medication whether prescribed or not (with the exception of contraceptives, including vitamins and herbal remedies such as St John's Wort.
* Subject has participated in a clinical study with a New Chemical Entity (NCE) within the past 3 months
* Infected with the Hepatitis B, Hepatitis C, or HIV virus
* Subject has a history of drug or other allergy, which, in the opinion of the Investigator, contraindicates their participation

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11-29 (Actual); Primary Completion 2008-01-08 (Actual); Study Completion 2008-01-08 (Actual)

PRIMARY OUTCOMES:
FEV1 at intervals | during the 10 week study
Cardiac monitoring at intervals | during the 10 week study

SECONDARY OUTCOMES:
Plasma concentrations of GSK961081 at intervals | during the 10 week study
PK parameters at intervals | during the 10week study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study MAB108115 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MAB108115?search=study&search_terms=MAB108115#rs
- Available data/document: Individual Participant Data Set: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MAB108115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register